CLINICAL TRIAL: NCT04058912
Title: RELATIONSHIP OF LOW-OVER RESERVE WITH PTEN-AKT-FOXO3 GENE EXPRESSION IN THE PRESENCE OF ENDOMETRIOMAS
Brief Title: PTEN-AKT-FOXO3 Gene Expression Relation With Low-ovarian Reserve in Endometriomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, : Principal Investigator. Professor, Obstetrician and Gynecologist, Uludag University
Other Study IDs: UU-MREC-2019-5/28
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Reserve, Endometrioma, PTEN-AKT-FOXO3 Gene Expression
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PATİENCE GROUP: 1. To be in the range of 18-40 years
  2. Patients with an operation indication with >=5 cm endometrioma
     1. Symptomatic patients due to endometrioma (dysmenorrhea, dyspareunia, chronic pelvic pain, etc.)
     2. Patients who will be followed for IVF cycle due to infertility
  Interventions: Genetic: PTEN-AKT-FOXO3 Gene Expression
- PATİENCE-CONTROL GROUP: 1. To be in the range of 18-40 years
  2. Patients with operation plan due to non-endometrioma ovarian pathologies
     1. Symptomatic patients with benign ovarian pathology (such as chronic pelvic pain, compression, syphilomas, dysmenorrhea, dyspareunia, etc.)
     2. Asymptomatic, despite a 6-month follow-up period, increase in cyst size or become symptomatic
  Interventions: Genetic: PTEN-AKT-FOXO3 Gene Expression

INTERVENTIONS:
Genetic: PTEN-AKT-FOXO3 Gene Expression — In the patient and patient control groups, 0.5 mm tissue strip will be removed for pathology from the cyst wall removed during surgery. and tissue samples will be stored in phosphate buffered saline at -80 C and PTEN-AKT-FOXO3 gene expression level will be evaluated by RT-PCR analysis.

SUMMARY:
In this study, we aimed to investigate the relationship between PTEN-AKT-FOXO3 gene expression and decrease in ovarian reserve in the presence of endometrioma and other benign ovarian pathologies.

DETAILED DESCRIPTION:
It is known that the presence of endometrioma negatively affects ovarian reserve. The development of endometriosis and the effect of the presence of endometrioma on ovarian reserve due to decreased PTEN expression are considered. This study was designed to compare ovarian PTEN-AKT-FOXO3 gene expression and ovarian reserve in patients with underwent surgery caused by endometrioma and those who had ovarian pathology due to other benign causes and PTEN-AKT-FOXO3 gene expression level will be evaluated by RT-PCR analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1) To be in the range of 18-40 years 2) Patients with an operation indication with >=5 cm endometrioma 3) Patients with operation plan due to non-endometrioma ovarian pathologies

Exclusion Criteria:

* 1)Patients over the age of 40 2)Patients with suspected malignancy 3)Follow-up patients without indications for operation

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The study population is the patients examined for ovarian endometriomas and other benign ovarian pathologies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-05-27 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
PTEN AKT FOXO3 gene expression | 30 minutes
  In the patient and patient control groups, 0.5 mm tissue strip will be removed for pathology from the cyst wall removed during surgery. and tissue samples will be stored in phosphate buffered saline at -80 C and PTEN-AKT-FOXO3 gene expression level will be evaluated by RT-PCR analysis.

CONTACTS AND LOCATIONS:
Overall Officials: GURKAN UNCU, Prof, Study Director — ULUDAG UNIVERSITY HOSPITAL BURSA TURKEY
Locations (1):
- Uludag University Hospital, Department of Obstetrics and Gynecology, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govatati S, Kodati VL, Deenadayal M, Chakravarty B, Shivaji S, Bhanoori M. Mutations in the PTEN tumor gene and risk of endometriosis: a case-control study. Hum Reprod. 2014 Feb;29(2):324-36. doi: 10.1093/humrep/det387. Epub 2013 Oct 23. PMID 24154570
- [Background] Kasapoglu I, Ata B, Uyaniklar O, Seyhan A, Orhan A, Yildiz Oguz S, Uncu G. Endometrioma-related reduction in ovarian reserve (ERROR): a prospective longitudinal study. Fertil Steril. 2018 Jul 1;110(1):122-127. doi: 10.1016/j.fertnstert.2018.03.015. Epub 2018 Jun 20. PMID 29935810